CLINICAL TRIAL: NCT05094050
Title: Parkinson's Disease: A Comparative Study of Levodopa and Carbidopa Bioavailability Following Foslevodopa/Foscarbidopa Infusion at Different Subcutaneous Sites in Parkinson's Disease Patients
Brief Title: Study to Assess How ABBV-951 is Absorbed When Administered at Different Subcutaneous Sites of Adult Participants With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20-339
Record Dates: First submitted 2021-10-20; First posted 2021-10-26 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Foslevodopa/foscarbidopa; ABBV-951; Levodopa (LD); Carbidopa (CD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: ABBV-951 (Experimental): Participants will receive ABBV-951 for 2 consecutive days in the abdomen (Period 1), flank (Period 2), arm (Period 3) and thigh (Period 4).
  Interventions: Drug: ABBV-951
- Arm 2: ABBV-951 (Experimental): Participants will receive ABBV-951 for 2 consecutive days in the arm (Period 1), abdomen (Period 2), thigh (Period 3) and flank (Period 4).
  Interventions: Drug: ABBV-951
- Arm 3: ABBV-951 (Experimental): Participants will receive ABBV-951 for 2 consecutive days in the thigh (Period 1), arm (Period 2), flank (Period 3) and abdomen (Period 4).
  Interventions: Drug: ABBV-951
- Arm 4: ABBV-951 (Experimental): Participants will receive ABBV-951 for 2 consecutive days in the flank (Period 1), thigh (Period 2), abdomen (Period 3) and arm (Period 4).
  Interventions: Drug: ABBV-951

INTERVENTIONS:
Drug: ABBV-951 — Continuous Subcutaneous Infusion (CSCI)
  Other Names: Foslevodopa/foscarbidopa

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which means it affects the brain. This study will evaluate how ABBV-951 is absorbed under the skin of participants with PD when administered to arm, thigh and flank compared to the abdomen.

ABBV-951 is an investigational drug being developed for the treatment of PD. Study doctors randomly assign participants to 1 of 4 groups, called treatment arms. Each treatment arm receives ABBV-951 administered in a different order in the arm, high, flank and abdomen. Approximately 12 adult participants over 30 years with a diagnosis of PD will be enrolled in approximately 10 sites in the United States.

Participants will receive continuous (24hours/day) subcutaneous infusion of ABBV-951 for 2 consecutive days for each infusion site (arm, thigh, flank and abdomen), for a total duration of treatment up to 12 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will be confined at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires. Adverse events will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease (PD) that is Levodopa-responsive.
* Must be taking a minimum of 400 mg/day of levodopa equivalents (LE) and be judged by the investigator to have motor symptoms inadequately controlled by current therapy.
* Must have recognizable/identifiable "Off" and "On" states (motor fluctuations), and have a minimum daily average of 2.5 hours of "Off" time (with a minimum of 2 hours of "Off" time each day).

Exclusion Criteria:

- History of significant skin conditions or disorders (e.g., psoriasis, atopic dermatitis, etc.) or evidence of recent sunburn, acne, scar tissue, tattoo, open wound, branding, or colorations that in the investigator's opinion would interfere with the infusion of the study drug or could interfere with study assessments.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Levodopa (LD) | Up to 8 Days
  Maximum observed plasma concentration (Cmax) of Levodopa (LD).
Area Under the Plasma Concentration-Time Curve (AUC) for the 24-hour Interval of LD | Up to 8 Days
  Area under the plasma concentration-time curve (AUC) for the 24-hour interval of LD.
Minimum Observed Plasma Concentration (Cmin) of LD | Up to 8 Days
  Minimum observed plasma concentration (Cmin) of LD.
Degree of Fluctuation (DFL) of LD | Up to 8 Days
  DFL = (Cmax-Cmin)/(average plasma concentration).
Swing of LD | Up to 8 Days
  Swing = (Cmax-Cmin)/Cmin.
Maximum Observed Plasma Concentration (Cmax) of Carbidopa (CD) | Up to 8 Days
  Maximum observed plasma concentration (Cmax) of CD.
Area Under the Plasma Concentration-Time Curve (AUC) for the 24-hour Interval of CD | Up to 8 Days
  Area under the plasma concentration-time curve (AUC) for the 24-hour interval of CD.
Minimum Observed Plasma Concentration (Cmin) of CD | Up to 8 Days
  Minimum observed plasma concentration (Cmin) of CD.
Degree of Fluctuation (DFL) of CD | Up to 8 Days
  DFL = (Cmax-Cmin)/(average plasma concentration).
Swing of CD | Up to 8 Days
  Swing = (Cmax-Cmin)/Cmin.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (10):
  - University of Colorado Hospital /ID# 229974, Aurora, Colorado
  - Georgetown University Hospital /ID# 230224, Washington D.C., District of Columbia
  - Rush University Medical Center /ID# 229983, Chicago, Illinois
  - Carolina Phase 1, LLC /ID# 239836, Raleigh, North Carolina
  - The Movement Disorder Clinic of Oklahoma /ID# 238610, Tulsa, Oklahoma
  - Vanderbilt University Medical Center /ID# 230255, Nashville, Tennessee
  - Parkinson Disease Movement Disorders Clinic /ID# 245791, Austin, Texas
  - Texas Movement Disorder Specialists /ID# 238607, Georgetown, Texas
  - Baylor College of Medicine - Baylor Medical Center /ID# 239631, Houston, Texas
  - University of Utah Health Care /ID# 241219, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No